CLINICAL TRIAL: NCT02991625
Title: Brain Imaging Study on Biomarkers for Chronic Back Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1021846
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebos (Experimental): Chronic Back Pain participants will enter an optional placebo trial. This phase of the study will test the clinical usefulness of the biomarkers. We will measure how expectation of starting a new treatment reduces 'clinical back pain' in each participant. Positive treatment expectations will be induced by giving them capsules containing inert material and telling them that the capsules contain an effective drug that has been approved for treating Chronic Back Pain. They will be requested to take two capsules twice a day and report their pain on paper forms organized as a calendar.
  Interventions: Other: Placebos
- Waitlist (Other): Chronic Back Pain participants will not be given any placebo and will be requested to report their pain on paper forms organized as a calendar.
  Interventions: Other: Waitlist
- Healthy Controls (Other): Healthy control participants will complete the main part of the study, but will not be asked to take a placebo or be placed on a waitlist.
  Interventions: Other: Healthy Controls

INTERVENTIONS:
Other: Placebos — Positive treatment expectations will be induced by giving participants capsules containing inert material and telling them that the capsules contain an effective drug that has been approved for treating Chronic Back Pain. They will be requested to take two capsules twice a day and report their pain on paper forms organized as a calendar.
  Arms: Placebos
Other: Waitlist — These Chronic Back Pain participants will not be given any placebos and will be requested to report their pain on paper forms organized as a calendar.
  Arms: Waitlist
Other: Healthy Controls — Healthy control participants will not receive a placebo drug or be put on a waitlist.
  Arms: Healthy Controls

SUMMARY:
The study proposes to investigate the factors related to a person that can enhance or reduce the effectiveness of pain treatments in people suffering with chronic pain. Treatment response to pain killers in a person may be related to their brain, genetics, social, and psychological makeup. The investigators aim to study these factors to identify and develop feasible and robust indicators based on a person's biological makeup (also called biomarkers).

DETAILED DESCRIPTION:
Drugs used for managing chronic pain have not proven to be effective and chronic pain continues to cost Canadians $60 billion a year without truly helping those who suffer. The study proposes to investigate the factors related to a person that can enhance or reduce the effectiveness of pain treatments in people suffering with chronic pain. Treatment response to pain killers in a person may be related to their brain, genetics, social, and psychological makeup. The investigators aim to study these factors to identify and develop feasible and robust indicators based on a person's biological makeup (also called biomarkers). These biomarkers will allow doctors and researchers to predict more accurately which treatment and prevention strategies for a particular disease will work in which groups of people. These measures will offer new opportunities for improving treatment such as by tailoring treatment to meet the specific needs of each patient based on his/her biological and psychological makeup. Towards the specific aim, data will first be collected in several experimental domains for studying treatment expectations (cognitive, psychosocial, brain-related, genetic). These 'experimental' data will be compared between chronic back pain (CBP) and healthy participants to yield new understanding of the factors that govern treatment response. At the end of experimental data collection, the investigators will collect data in the 'clinical' domain. Hence, at the end of the experimental sessions, a subset of CBP participants will receive a mock drug (placebo disguised as an approved pain treatment) and another subset will provide pain ratings only and hence serve as a waiting list control for the placebo trial. Data will be studied in steps to understand factors that mediate treatment outcomes and finally the investigators will use advanced computational tools used for big data analysis and aim to identify factors that can be used as biomarkers and precision medicine tools.

ELIGIBILITY:
Inclusion Criteria:

Chronic pain participant inclusion criteria:

1. 18-75 years of age
2. Right-handed
3. Meet the classification criteria of chronic low back pain (having low back pain for more than 6 months), as determined by a physician and documented in the participant's medical record.
4. At least 4/10 clinical pain on the Brief Pain Inventory Scale on average during the two weeks prior to enrollment
5. Comfortable completing (reading and writing) questionnaires and tasks with English language instructions

Healthy participant inclusion criteria:

1. 18 - 75 years of age
2. Right-handed
3. Comfortable completing (reading and writing) questionnaires and tasks with English language instructions

Exclusion Criteria:

Chronic pain participant exclusion criteria:

1. History of cardiac, respiratory, or nervous system disease that may interfere with participation in the study or cause heightened potential for adverse outcome. For example: asthma or claustrophobia
2. Presence of any contraindications to MRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy

Healthy participant exclusion criteria:

1. Acute or chronic pain
2. History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment and by asking the participant about their comfort level and ability, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma or claustrophobia
3. Presence of any contraindications to MRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Pain modulation - using an experimental task that tests a person's ability to form positive expectations | 3 days after first visit
  Brain imaging will be used to assess each participant's capacity to endogenously adjust pain perception with changes in expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Javeria A Hashmi, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Nova Scotia Health Authoity QEII, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hashmi JA, Baliki MN, Huang L, Baria AT, Torbey S, Hermann KM, Schnitzer TJ, Apkarian AV. Shape shifting pain: chronification of back pain shifts brain representation from nociceptive to emotional circuits. Brain. 2013 Sep;136(Pt 9):2751-68. doi: 10.1093/brain/awt211. PMID 23983029
- [Background] Vase L, Vollert J, Finnerup NB, Miao X, Atkinson G, Marshall S, Nemeth R, Lange B, Liss C, Price DD, Maier C, Jensen TS, Segerdahl M. Predictors of the placebo analgesia response in randomized controlled trials of chronic pain: a meta-analysis of the individual data from nine industrially sponsored trials. Pain. 2015 Sep;156(9):1795-1802. doi: 10.1097/j.pain.0000000000000217. PMID 25955965
- [Background] Hashmi JA, Kong J, Spaeth R, Khan S, Kaptchuk TJ, Gollub RL. Functional network architecture predicts psychologically mediated analgesia related to treatment in chronic knee pain patients. J Neurosci. 2014 Mar 12;34(11):3924-36. doi: 10.1523/JNEUROSCI.3155-13.2014. PMID 24623770
- [Background] Hashmi JA, Baria AT, Baliki MN, Huang L, Schnitzer TJ, Apkarian VA. Brain networks predicting placebo analgesia in a clinical trial for chronic back pain. Pain. 2012 Dec;153(12):2393-2402. doi: 10.1016/j.pain.2012.08.008. Epub 2012 Sep 15. PMID 22985900
- [Derived] Sunavsky A, Hashmi MA, Robertson JW, Veinot J, Hashmi JA. The nucleus accumbens-prefrontal connectivity as a predictor of chronic low back pain. Pain. 2025 Oct 1;166(10):e363-e377. doi: 10.1097/j.pain.0000000000003620. Epub 2025 May 15. PMID 40388641